CLINICAL TRIAL: NCT03008265
Title: Just a Fascial Dehiscence? Nationwide Cohort Study on the Mortality Associated With Fascial Dehiscence After Colonic Resection
Brief Title: Fascial Dehiscence and Mortality
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kristian Kiim Jensen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kiim Jensen, Dr., Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: 2016-Fascial-dehiscence-mort
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Wound Breakdown
Keywords: Fascial dehiscence; Mortality
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Colonic cancer resection
  Interventions: Other: Postoperative fascial dehiscence

INTERVENTIONS:
Other: Postoperative fascial dehiscence

SUMMARY:
Nationwide cohort study on short- and long-term mortality of patients with and without postoperative fascial dehiscence.

The cohort will be comprised of patient undergoing open colonic resection for colonic cancer registered in the Danish Colorectal Cancer Group Database. The exposure is fascial dehiscence and the outcome of interest 30-day, 3- and 5-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent open colonic resection identified in the DCCG

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent open colonic resection for carcinoma in the period 2001-2008 in Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
3-year mortality | Three years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Jensen, MD, Principal Investigator — Digestive Disease Center, Bispebjerg Hospital
Locations (1):
- Digestive Disease Center, Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided